CLINICAL TRIAL: NCT01318239
Title: Study of Perfusion and Diffusion Magnetic Resonance Imaging, and Phosphorylation of Circulation Endothelial Cells to Determine Anti-angiogenic Effect in Patients With Colorectal Liver Metastasis in Chemotherapeutic Regimens Including Avastin
Brief Title: Perfusion and Diffusion Magnetic Resonance Imaging, and Phosphorylation of Circulation Endothelial Cells to Determine Anti-anogenic Effect of Chemotherapeutic Regimens in Colorectal Liver Metastasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2010-0047
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Chemotherapy with Avastin (Experimental)
  Interventions: Procedure: DCE MRI
- Standard Chemotherapy only (Active Comparator)
  Interventions: Procedure: DCE MRI

INTERVENTIONS:
Procedure: DCE MRI — MRI and blood test(VEGFR2 signaling assay) will be undergoing at three time points in the patients with Avastin chemotherapy; at baseline (pretreatment), 3 days after Avastin alone treatment, 3 days after Avastin combined chemotherapy (about 10 days after initial Avastin alone treatment).
  MRI and blood test(VEGFR2 signaling assay) will be undergoing at two time points in the patients who will get chemotherapy without antiangiogenic agent; at baseline (pretreatment), 3 days after chemotherapy.

SUMMARY:
The purpose of our study is to establish the accuracy of the perfusion MRI parameters and the availability of the VEGFR2 signaling assay using phosphospecific flow cytometry in predicting the response of liver metastasis from colorectal cancer to treatment with antiangiogenic agent.

DETAILED DESCRIPTION:
The purpose of our study is to establish the accuracy of the perfusion MRI parameters and the availability of the VEGFR2 signaling assay using phosphospecific flow cytometry in predicting the response of liver metastasis from colorectal cancer to treatment with antiangiogenic agent.

IRB approval will be obtained to enroll 60 naïve patients (30 patients who will get antiangiogenic agent (Avastin) combined chemotherapy and 30 patients who will get chemotherapy without antiangiogenic agent) with liver metastasis from colorectal cancer. MRI and blood test (VEGFR2 signaling assay) will be undergoing at three time points in the patients with Avastin chemotherapy; at baseline (pretreatment), 3 days after Avastin alone treatment, 3 days after Avastin combined chemotherapy (about 10 days after initial Avastin alone treatment). MRI and blood test (VEGFR2 signaling assay) will be undergoing at two time points in the patients who will get chemotherapy without antiangiogenic agent; at baseline (pretreatment), 3 days after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have single or multiple liver metastasis from colorectal cancer
* Patients willing to undergo the study procedure
* Patients who are fully informed about the study and have signed the informed consent form
* 60 patients (30 patients who will get antiangiogenic agent(Avastin) combined chemotherapy and 30 patients who will get chemotherapy without antiangiogenic agent)

Exclusion Criteria:

* Patients (men or women) under 20 years of age
* Patients who have previously entered this study
* Patients who have received or will receive any investigational drug 48 hours before injection of the study drug or during study participation
* Women who are pregnant, lactating or who are of childbearing potential and have not had a negative pregnancy test at baseline visit
* Patients not eligible to contrast media injection according to product labeling
* Patients with a contraindication for MRI or CT
* Patients with impaired renal function (e.g. acute renal failure) or patients on dialysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
MR perfusion parameter | 3 days after administrating avastin
  MR perfusion parameter(Ktrans, Kep, Ve)

SECONDARY OUTCOMES:
diffusion parameter | 3 days after an anti-cancer medicine
  diffusion parameter(ADC; apparent diffusion coefficient)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea